CLINICAL TRIAL: NCT00753636
Title: Phase II Safety and Tolerability of Isradipine (A Potential Neuroprotective Agent) in Patients With Parkinson's Disease- Stage II
Brief Title: Parkinson's Disease Isradipine Safety Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: Northwestern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Tanya Simuni, Professor of Neurology, Northwestern University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Isradipine II
Record Dates: First submitted 2008-09-13; First posted 2008-09-16 (Estimated); Results first posted 2011-07-01 (Estimated); Last update posted 2021-11-15 (Actual); Status verified 2021-11

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Isradipine; Neuroprotection
MeSH Terms: conditions — Parkinson Disease | interventions — Isradipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dynacirc CR (Isradipine) (Experimental): Dynacirc CR (Isradipine) will start at 5mg dose and increased in increments of 5mg every 2 weeks
  Interventions: Drug: Dynacirc CR (Isradipine)

INTERVENTIONS:
Drug: Dynacirc CR (Isradipine) — Dynacirc CR is given by the recommended schedule for titration. Subjects start on a 5mg dose and are increased in increments of 5mg every 2 weeks provided that the subjects do not have significant adverse events or symptomatic orthostatic hypotension.
  Other Names: Isradipine

SUMMARY:
The objective of this study is to establish the safety and tolerability of isradipine, sustained release preparation in patients with PD. This study is a logical continuation of the project that is being completed now and is conducted in preparation to NIH submission of the pivotal study on the efficacy of this agent for neuroprotection in PD. This study is conducted in parallel with Dr. Surmeier's work on further development of the preclinical data. The focus of his work now is to establishing the correlation between the dose that demonstrated neuroprotective effect in animal model and the dose used for clinical practice.

Hypothesis 1: Patients with PD will be able to tolerate isradipine across the FDA recommended dose range. We expect 10% attrition due to hypotensive effect of the agent.

Hypothesis 2: Patients with PD and concomitant stable hypertension will be able to tolerate isradipine provided that the dose of the concomitant antihypertensive agent is adjusted based on the blood pressure reading.

DETAILED DESCRIPTION:
Isradipine safety profile Isradipine, FDA approved for treatment of hypertension since 1990, has a well established data on its efficacy and safety in the hypertensive population (see package insert, Appendix 3). The side effect profile of isradipine is related to the primary mechanism of action of the agent as a vasodilator of the vascular smooth muscles and myocardium, and includes hypotension, bradycardia, weakness, and syncope. As per package insert, the most common adverse effects are headache (13.7% with active treatment versus 14% placebo), dizziness (7.3 vs 4.4) and peripheral edema as reflection of the vasodilatory effect which is dose dependent with incidence of about 3.5% at 5 mg, 8.7% at 10 mg and 8.5% at 20 mg. Of note the incidence of edema is substantially lower compared to CR preparation (9:13:36% for the respective doses). The other side effects include angina, asthenia, flushing, heart failure, and palpitations. According to the package insert, the adverse effects are usually not serious, dose dependent, and respond well to dose reduction or discontinuation of therapy. Isradipine has no effect on atrioventricular or sinoatrial conduction. The only absolute contraindications for isradipine are hypersensitivity to DHP compounds and hypotension defined as systolic blood pressure below 90 mm Hg. Until our studies, isradipine has not been tested in the PD population.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with idiopathic Parkinson's disease age 30-75
2. Hoehn and Yahr stage <2.5
3. PD duration less than 5 years
4. For the subjects treated with PD medications, the regimen has to be stable for >1 month prior to enrollment

Exclusion Criteria:

1. Atypical Parkinsonian syndrome
2. Patients with history of stable hypertension treated with other antihypertensive agents will be allowed provided that the doses of concomitant anti HTN therapy can be reduced/adjusted during the study based on the BP readings. The number of concomitant antihypertensive agents should not exceed two. The dose of concomitant antihypertensive agents has to be stable for > 1 month
3. Presence of orthostatic hypotension at the screening visit defined as > 20 mmHg change in systolic BP and 10mm change in diastolic BP after 2 min of standing, or baseline BP <90/60.
4. Presence of other medical conditions that in the opinion of the investigator will preclude safe use of the drug.
5. Presence of cognitive dysfunction as determined by MMSE score <24
6. Failure to sign the informed consent
7. Inability to cooperate with the study procedures
8. Presence of motor fluctuations
9. History of bradycardia defined as heart rate < 55
10. Women of childbearing potential who are not surgically sterilized have to use a reliable measure of contraception and have a negative urine pregnancy test at screening
11. Participation in other investigational drug trials within 30 days prior to screening
12. History of brain surgery for Parkinson's Disease.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2008-04; Primary Completion 2009-06 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Simuni, M.D., Principal Investigator — Northwestern University
Locations (1):
- 710 N. Lake Shore Dr., Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 35 Screened
Period: Overall Study
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Started | 31
Completed | 25
Not Completed | 6

BASELINE CHARACTERISTICS:
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.87 (8.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 31

OUTCOME MEASURES:

1. Primary Outcome: Tolerability of Isradipine Based on the Number of Participants That Complete the Study
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Participants | 25

2. Secondary Outcome: Safety of the Standard Titration Schedule in PD Population as Measured by the Number of Patients That Are Able to Increase the Dose to 20 mg Daily
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Participants | 16

3. Secondary Outcome: Number of Participants That Tolerated Each Dose of Isradipine
Description: Tolerability= maximum tolerated dose
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Participants
  20mg | 16
  15mg | 5
  10mg | 6
  5mg | 4

4. Secondary Outcome: Number of Participants That Tolerated Each Dose Level of Isradipine Between PD Patients Treated With Antihypertensive Agent and Not on Antihypertensive Agent
Description: At the time of enrollment, some patients were currently being treated with antihypertensive agents including Propanolol, Toprol, Lisinopril, Diovan, Norvasc.
  HTN+: Participants on an antihypertensive agent HTN-: Participants not on an antihypertensive agent
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Participants
  HTN+ 20mg | 2
  HTN+ 15mg | 3
  HTN+ 10 mg | 1
  HTN+ 5mg | 0
  HTN- 20mg | 14
  HTN- 15mg | 2
  HTN- 10mg | 5
  HTN- 5mg | 4

5. Secondary Outcome: Number of Participants That Completed the Study at Each Dose Level of Isradipine
Time Frame: 1 year
Measure: Number; unit: Participants
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
Participants
  20mg | 16
  15mg | 4
  10mg | 4
  5mg | 1

6. Secondary Outcome: Change in Motor UPDRS Scores: Baseline vs. Final Visit
Description: Baseline visit = Week 0 Final visit = Week 12
  Unified Parkinson's Disease Rating Scale (UPDRS)is made up of the following sections:
  Part I: evaluation of Mentation, behavior, and mood Part II: self evaluation of the activities of daily life Part III: clinician-scored motor evaluation Part IV: Hoehn and Yahr stating of severity of Parkinson disease. Part V: Schwab and England ADL scale Only part three was used for this assessment.
  The higher the UPDRS score, the greater the disability from PD.
  The range for scores for Section III is 0 to 108.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: UPDRS Part III Score
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
UPDRS Part III Score
  Baseline | 7.61 (3.01)
  Final | 7.08 (2.68)

7. Secondary Outcome: Pharmacokinetic Data - Mean Serum Concentration and Dosage Exposure Across the Dose Range of Isradipine
Description: Mean Plasma Concentration (+/- SD ng/mL)
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Number analyzed (Participants) | 31
ng/mL
  20 mg | 2.48 (1.16)
  15 mg | 2.53 (1.33)
  10 mg | 1.53 (0.72)
  5 mg | 0.68 (0.38)

ADVERSE EVENTS:
Groups:
- Isradipine 20mg, 15mg, 10mg or 5 mg: A group is defined by the highest dose received by the subject. Subjects are started at 5mg dose, and may end at the highest dose of 20mg, depending on how they tolerate the drug. Thus, assignment to a group is not randomized but relies on the last/highest dose received.
Arm/Group | Isradipine 20mg, 15mg, 10mg or 5 mg
Serious Adverse Events (participants affected / at risk) | 0/31
Other Adverse Events (participants affected / at risk) | 31/31
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Isradipine 20mg, 15mg, 10mg or 5 mg (N=31)
Leg Edema (Musculoskeletal and connective tissue disorders) | 17 (17)
Fatigue (General disorders) | 9 (9)
Dizziness (General disorders) | 10 (10)
Headache (General disorders) | 5 (5)
Nausea (General disorders) | 5 (5)
Cough (General disorders) | 2 (2)
Soar Throat (General disorders) | 2 (2)
Sinuses (General disorders) | 2 (2)
Shortness of breath (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erectile/sexual Dysfunction (Reproductive system and breast disorders) | 2 (2)
Cold (General disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No